CLINICAL TRIAL: NCT06574607
Title: Effects of a Contextual Decision-making Learning Materials on Nurses in Two Years Learning Performance for Abdominal and Pelvic Traumatic Severe Bleeding Care
Brief Title: Effects of a Contextual Decision-making Materials on Junior Nurses in Traumatic Learning Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202304128RIND
Record Dates: First submitted 2023-11-26; First posted 2024-08-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-08

CONDITIONS: Abdominal Injury; Pelvic Injury
Keywords: Decision Guidance; Care of Severe Bleeding in Abdominal-Pelvic Trauma; Scenario-Based Learning; Two-Year Registered Nursing; Clinical Reasoning Assessment; Abdominal injury; Pelvic Injury
MeSH Terms: conditions — Abdominal Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Device: Interactive Educational Material for Decision-Making
- control group (Active Comparator)
  Interventions: Device: Interactive Educational Material

INTERVENTIONS:
Device: Interactive Educational Material for Decision-Making — Using severe bleeding from abdominal-pelvic trauma as a scenario case, implementing decision-making teaching strategies to guide learners, and examining the intervention through this research
  Arms: experimental group
Device: Interactive Educational Material — Teaching with scenario-based interactive materials without incorporating any teaching strategies
  Arms: control group

SUMMARY:
Trauma leading to severe bleeding is one of the reasons for the high mortality rate in trauma patients, resulting in multiple and complex injuries from various accidental mechanisms. However, patients with abdominal-pelvic trauma accidents rank among the top three common accidents in the emergency department. There is a potential for both trauma and severe internal bleeding, making the care of such patients even more challenging. Currently, trauma nursing education focuses on emergency medical care, and teaching on the care of abdominal-pelvic trauma occupies only a small part of the entire nursing curriculum.

In addition to insufficient knowledge teaching in emergency trauma medical care, learning relies heavily on the arrangement of clinical internships, and obtaining practical experience in the care of abdominal-pelvic trauma is often difficult. In the current era of thriving digital learning, allowing learning to be more diverse and unrestricted by time and location, it is essential to integrate appropriate guiding strategies alongside digital technology to make learning more efficient and promote meaningful learning.

Therefore, this study introduces decision trees into an interactive scenario-based learning environment for the care of severe bleeding due to abdominal-pelvic trauma. The decision tree is coupled with a decision-making strategy, utilizing the relationships between leaf nodes to guide learners in clarifying their misconceptions, ultimately leading them to make appropriate decisions to reach the final nodes and solve problems.

To understand the effectiveness of this study, a real experimental research design is adopted to investigate the impact of introducing decision tree-based interactive teaching materials on the care of severe bleeding in abdominal-pelvic trauma situations on the professional knowledge, self-efficacy, clinical reasoning assessment ability, and technology acceptance of surgical nursing students over a two-year period. It is hoped that this interactive teaching material for the care of severe bleeding in abdominal-pelvic trauma scenarios will enhance learners' professional knowledge, self-efficacy, clinical reasoning assessment, and technology acceptanc.

ELIGIBILITY:
Inclusion Criteria:

* Holding a nursing license, employed, and having job registration in the same institution.
* Those who are willing to participate in this study, are informed, and have provided consent by signing the informed consent form

Exclusion Criteria:

* Those who have completed a service period of more than two years
* Those who refuse to participate in this study.
* Non-Surgical Department ward nurses

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
The effect of "Interactive Educational Material for Decision-Making"intervention program on Abdominal and Pelvic Traumatic Severe Bleeding care knowledge learning outcome | up to 1 month
  TThe changes of Questionnaire score of Abdominal and Pelvic Traumatic Severe Bleeding care knowledge, Questionnaire including:
  Abdominal and Pelvic Traumatic Severe Bleeding knowledge Scores range from 0 to 15, with higher scores representing higher knowledge of Abdominal and Pelvic Traumatic Severe Bleeding care
The effect of "Interactive Educational Material for Decision-Making"intervention program on Abdominal and Pelvic Traumatic Severe Bleeding care Technology Acceptance learning outcome | up to 1 month
  The changes of Questionnaire score of Abdominal and Pelvic Traumatic Severe Bleeding care Technology Acceptance, Questionnaire including:
  Technology Acceptance Scale:Scores range from 1 to 5, with higher scores representing better Technology Acceptance.
The effect of "Interactive Educational Material for Decision-Making"intervention program on Abdominal and Pelvic Traumatic Severe Bleeding care Clinical Reasoning Evaluation Simulation learning outcome | up to 1 month
  The changes of Questionnaire score of Abdominal and Pelvic Traumatic Severe Bleeding care Clinical Reasoning Evaluation Simulation , Questionnaire including:
  Clinical Reasoning Evaluation Simulation Tool(CREST): Scores range from 0 to 100, with higher scores representing more positive Clinical Reasoning Evaluation beliefs.
The effect of "Interactive Educational Material for Decision-Making"intervention program on Abdominal and Pelvic Traumatic Severe Bleeding care self-efficacy learning outcome | up to 1 month
  The changes of Questionnaire score of Abdominal and Pelvic Traumatic Severe Bleeding care self-efficacy will be measured, Questionnaire including:
  Self-Efficacy Scale:Scores range from 1 to 5, with higher scores representing better self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No